CLINICAL TRIAL: NCT07377799
Title: PRospective Cohort Study for the Identification of Subclinical Atrial Fibrillation In Patients With Significant Primary Mitral Valve Regurgitation
Brief Title: Study for the Identification of Subclinical Atrial Fibrillation In Patients With Significant Primary Mitral Regurgitation
Acronym: PRIME-LOOP
Status: Not yet recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lauge Østergaard, PRospective cohort study for the Identification of Subclinical atrial fibrillation In patients with significant primary Mitral valve regurgitation, Rigshospitalet, Denmark
Other Study IDs: 16-0302-9; NNF23OC0081668 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Mitral Regurgitation; Atrial Fibrillation (AF)
Keywords: degenerative mitral regurgitation; asymptomatic; atrial fibrillation; subclinical atrial fibrillation
MeSH Terms: conditions — Mitral Valve Insufficiency; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ILR

SUMMARY:
The PRIME-LOOP study is a prospective cohort investigating the burden of atrial fibrillation (AF) and subclinical AF in patients with moderate-severe or severe primary mitral regurgitation (MR). The study will use long-term cardiac monitoring with an implantable loop recorder (ILR) for up to three years to identify the burden of AF. Further, the study aims to examine the associated risk of adverse events among patients with detected AF as compared with patients without AF. Only patients with no or mild symptoms related to MR and without a class I indication for surgical intervention will be included. The study aims to include 100 patients.

Patients will be screened from the PRIME cohort - a prospective cohort of patients with primary MR in East Denmark.

DETAILED DESCRIPTION:
Purpose

There are two main purposes of this study: 1) to assess atrial fibrillation (AF) burden in patients with asymptomatic severe primary degenerative mitral regurgitation (MR) but no known AF using the CE marked Reveal LINQ™ Insertable Cardiac Monitor (ICM), and 2) to examine the association between subclinical AF and deterioration of left ventricular (LV) dysfunction, progression of symptoms, and time to surgery.

We hypothesize that:

1. Within one year of follow-up, up to 30% of patients with significant, asymptomatic, primary MR will have previously unknown AF detected when evaluated by continuous monitoring.
2. The deterioration of LV dysfunction, progression of symptoms, and time to surgery are aggravated by subclinical AF.

Background

Mitral regurgitation and atrial fibrillation MR is the second most common reason for heart valve surgery in the Western World and the most common valvular heart disease. For patients with severe primary MR the only curative approach is an invasive assessment, usually with mitral valve surgery. There exist clear guidelines for the assessment of patients with symptomatic severe primary MR and with a class I recommendation, surgery is recommended, level of evidence B. The evidence supporting this recommendation is based on observational data. However, timing of surgery is much debated, and no randomized controlled trials have been conducted, for the assessment of patients with asymptomatic severe primary MR. It has been of interest to identify factors associated with worse outcomes in this patient population in order to guide clinical decision of early surgery. AF is a common complication in patients with severe primary MR. Increased left atrial pressure from primary MR leading to left atrial enlargement and remodeling is hypothesized to be the pathophysiologic driver for the development of AF. From non-continuous electrocardiography (ECG) monitored patients, the incidence rate of AF has been around 20% within a 5 year period, however this study was conducted between 1989 and 1994 where monitoring devices were not as extensively used as in contemporary health care systems in the Western world.7 Another study identified AF among 32% of patients at the time of the primary MR diagnosis.8 Several observational studies have linked AF with worse outcomes, as compared with patients without AF - regardless of surgery. These observational findings have led to the guideline recommendation that patients with asymptomatic severe primary MR and AF should be considered for surgery (class IIa recommendation, level of evidence B). Studies investigating the interplay between AF and primary MR have primarily been limited by the absence of a clearly defined protocol for the detection of AF. Most commonly, AF was identified with an electrocardiogram taken concomitantly with the diagnostic echocardiography or at the discretion of the clinician following primary MR diagnosis. Compared with external loop recording, where patients are monitored continuously for 30 days, long-term continuous monitoring using an implantable loop recorder (ILR) has an up to three times higher rate for the detection of AF within one year in patients with ischemic stroke. Continuous heart rhythm monitoring and the detection of subclinical AF is being used more and more common, however which clinical consequences to draw from this finding is unknown in patients with severe MR. In cases of severe asymptomatic primary MR, where the identification of AF could influence the decision for surgery, employing a systematic and ongoing screening approach may aid in determining, whether AF is a factor associated with adverse outcomes. Additionally, this approach would provide insights into establishing the optimal time threshold for associating AF with worse outcomes.

Implantable loop recorder The Reveal LINQ insertable cardiac monitor or implantable loop recorder is a widely used device for detecting cardiac arrhythmias including AF. The insertion procedure is minimally invasive and requires little time and clinical resources. The device is placed under the skin of the chest and automatically records and remotely transmits arrhythmia episodes along with daily summary-level heart rhythm data to the clinician. Thresholds for arrhythmia annotation can be adjusted to accommodate the individual setting but have generally proven to have a very high sensitivity and high specificity for AF. Symptom-prompted ECG recordings can be transmitted by the use of a hand-held "symptom button" (Patient Assistant, PA96000) that comes with the device.15, 16 Additional remote transmissions to save all ECG material can be performed by the patient. The device has a battery-life of at least 3 years.

Methods

Design The study is designed as a case study with follow-up, involving 100 participants with asymptomatic or mildly symptomatic, moderate-severe or severe primary MR where surgical intervention is not planned. Participants will be screened for inclusion (see chapter 8) and upon study eligibility and consent from the participant, an ILR will be implanted. Participants will be screened from an already established prospective cohort of patients with primary MR (The PRIME cohort, p-2025-18689). Patients included in this cohort have already consented to be contacted for enrolment in studies related to primary MR. Hence, inclusion will not rely on screening in the clinic.

From the day of implantation, the burden of AF will be remotely monitored. When data on AF burden has been collected, the impact of AF burden on clinical outcomes will be examined.

Trial specific treatment/evaluations Participating in this trial, requires the participantto meet at Rigshospitalet for a total of three site visits: at baseline, after 12 months and after 36 months. On the first visit, the participant will have the ILR implanted, participate in a medical interview, undergo echocardiography, blood tests, and the HeartQol questionnaire. The second visit will only include echocardiography, blood tests, and the HeartQol questionnaire, while the final visit will also include ILR explantation. The dates of visit will, if possible, be coordinated with the participant'sstandard consultation for primary MR, to minimize unnecessary time and travel costs for the participants.

Procedures upon detection of clinically relevant arrythmias During the three-year heart rhythm monitoring, potential arrythmias may be detected. If an arrhythmia is detected by the ILR, the coordinating investigator or a delegate will review the recorded rhythm via the CareLink® Remote Monitoring Network within one week of the alarm. Upon diagnostic uncertainty, data will be further reviewed by a senior cardiologist with expertise in arrythmia. If there is discrepancy in the assessment of the rhythm recorded by the ILR, a third senior cardiologist will independently evaluate the rhythm where at least two cardiologists are needed to confirm the diagnosis. All event data will be continuously logged in RedCap.

The following findings from the ILR will lead to participant contact and consideration of alterations in medical treatment:

1. A new AF episode ≥24 hours and a CHADS-VA score >1 will lead to participant contact and recommendation of oral anticoagulant treatment taking bleeding risk into account.

   Rate control will be considered with beta blocker, digoxin, or non-dihydropyridine calcium antagonist. Follow-up will be ensured to be at the general physician or the local department of cardiology.
2. Clinically significant bradyarrhythmia (i.e., 2nd degree atrioventricular block type 2 and complete heart block with ≥4 beats at rate <30 beats/min, sinus arrest/asystole >3 seconds) will lead to participant contact to identify symptoms such as syncope, shortness of breath, dizziness. A senior colleague and/or senior consultant, with specialty within cardiac pacemakers will be consulted for consideration of permanent pacemaker implantation.
3. Ventricular tachycardia (VT). The participant will be contacted in case of non-sustained or sustained VT to identify symptoms such as palpitations, chest pain, syncope, dizziness. In case of sustained VT, the participant will be admitted to the local cardiology award for consideration of an Implantable electronic device. In case of non-sustained VT referral to the local department of cardiology will be considered for non-invasive test for myocardial ischemia and consideration of initiation of beta blocker.

Alterations in medical treatment are warranted when one of the abovementioned findings may be identified to reduce the risk of ischemic stroke, heart failure, syncope, myocardial ischemia, cardiac arrest and can be prevented if timely and correct medical therapy is initiated.

The coordinating investigators will review alerts from the ILR and upon detection of one the abovementioned findings, alterations in medical management will be discussed with the principle investigator and the expert committee. The final decision as to whether trial participant will be informed of a secondary finding shall be made by the principal investigator, based on a clinical and ethical assessment and in accordance with applicable ethical guidelines and recommendations from the relevant ethics committee.

Procedures upon detection of other significant clinical findings Through blood tests and echocardiography, study personnel may identify previously undiagnosed conditions requiring further monitoring, diagnostic evaluation, or treatment initiation. If such findings occur, the participant will be informed and advised to contact their attending physician. As with arrhythmia detection, any subsequent interventions will be at the discretion of the partipant's attending physician.

Outcomes

The outcomes are examined during the three years from ILR implantation to ILR explantation. In addition, follow-up studies will be conducted at 5 and 10 years after explantation to further investigate the association between subclinical AF and adverse outcomes assessed from medical records. All outcomes are listed below.

Primary outcome Atrial fibrillation detection: Episode of ≥6 minutes of consecutive AF at any time during the 3-year monitoring time

Statistical considerations and data analyses

Statistical considerations The study is explorative in character, as the burden of AF in this population has not been examined with continuous monitoring previously. The expected proportion of participants that will be identified with AF, and the potential association with adverse outcomes, is based on pathophysiological theory and previous observational studies. In the LOOP-study, an ILR was assigned to 1,501 participants with no history of AF (median age 75 years) and at least one stroke risk factor (i.e., hypertension, diabetes, previous stroke, or heart failure).20 Among these, the authors found AF with a ≥6 min duration among 21% within 12 months and 31.8% within a median follow-up time of 39 months. With the considerable risk of AF linked to the presence of severe MR, we find it plausible that a similar or even higher rate of AF may be detected, as compared with that of the LOOP-study. Thus, we expect that this study will identify AF in up to 30% of the included participants within 12 months and 50% within 36 months. This rate is further supported by older studies that have identified AF in 20-30% of non-continuously monitored patients at the time of MR diagnosis. A key parameter in the clinical decision for surgical intervention is left ventricular end systolic diameter (LVESD). Patients with LVESD ≥40 mm have been associated with high mortality,21 hence LVESD ≥40 mm has become a class I indication for surgical intervention.2 We estimate that participants without AF detected by the ILR will have a mean LVESD of 35 mm with a standard deviation of 8 mm as measured by echocardiography at end of follow-up. For participants with AF as detected by ILR, the mean LVESD will be estimated at 40 mm. Assuming a two-sided alpha of 0.05 and a statistical power of 80% to detect this 5 mm increment in LVESD, a sample size of 40 participants per group is required for the study. Encountering dropouts and insecurity in estimates, we aim to enroll a total of 100 participants in total where it is estimated that around 50% will be categorized in the AF group and 50% will be categorized in the no AF group.

Data analyses This study will include 100 participants, all with an ILR. Should any dropouts occur, they will be replenished with new participants until the predetermined sample size is attained.

Secondary per-protocol analyses will be conducted, including only participants who complete the planned follow-up without major protocol deviations. The main analyses will be performed using multivariable Cox regression, assessing both the presence of AF as a baseline exposure and the occurrence of AF as a time-dependent covariate.

Participants who become pregnant during the study will be excluded from further monitoring from the date of pregnancy detection and censored at that time in the per-protocol analysis. Missing data will be handled using appropriate statistical methods depending on the extent and pattern of missingness (e.g., multiple imputation if data are missing at random).

Study participants

Eligible participants Participants eligible for inclusion are participants who are potential candidates for mitral valve surgery but do not meet the criteria for class I intervention and have not been diagnosed with AF, see below.

Inclusion criteria Asymptomatic/mildly symptomatic*, significant primary MR** LVEF ≥60% Native mitral valve Age ≥18 years old

Exclusion criteria Planned for mitral valve surgery LVESD ≥ 40 mm Prescence of cardiac pacemaker, ICD, cardiac resynchronization device, loop recorder, or a clinical indication for loop recorder Life expectancy < 1 year Pregnancy or lactating Prior diagnosis of AF

* Asymptomatic is defined as not being restricted in everyday activities due to dyspnea and have the functional capacity of walking to the second floor without being dyspneic (METS≥4). The evaluation of symptoms will be on the discretion of the treating physician.

**MR may be defined by either of two:

1. EROA ≥30 mm2 or regurgitation volume ≥45 mL.
2. If two cardiologists specialized in valvular heart assessment both consider the regurgitation to be moderate-severe or severe.

Abbreviations: MR: mitral regurgitation; AF: atrial fibrillation; ICD: implantable cardioverter defibrillator; LVESD: left ventricular end-systolic diameter; LVEF: left ventricular ejection fraction.

Discontinuation Participants reserve the right to terminate their involvement in the trial at any time. For participants who may become pregnant or is planned for cardiac valve surgery during the study period, the participant is informed to contact the coordinating investigator to have the ILR explanted. Likewise, investigators retain the authority to cease a participant's engagement if medical circumstances arise that preclude continued participation. In the event of discontinuation, all data pertaining to the participant will be retained up to the point of their withdrawal from the trial.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic/mildly symptomatic*, significant primary MR**
* LVEF ≥60%
* Native mitral valve
* Age ≥18 years old

Exclusion Criteria:

* Prior diagnosis of AF
* Prescence of cardiac pacemaker, ICD, cardiac resynchronization device, loop recorder, or a clinical indication for loop recorder
* LVESD ≥ 40 mm
* Planned for mitral valve surgery
* Life expectancy < 1 year
* Pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderat-severe or severe primary mitral regurgitation with no or mild symptoms without a class I indication for surgical intervention
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation detection | 3 years
  Episode of ≥6 minutes of consecutive AF at any time during the 3-year monitoring time

SECONDARY OUTCOMES:
Atrial fibrillation detection | 3 years
  Episode of ≥2 minutes of consecutive AF
Supraventricular tachycardia | 3 years
  Rate >150 bpm lasting ≥16 beats
Sinus arrest/asystole | 3 years
  Pauses > 3 seconds
Atrioventricular block | 3 years
  Second-degree or complete block with ≥4 beats at a rate <30 bpm
Sustained ventricular tachycardia | 3 years
  Rate >150 bpm lasting ≥30 seconds
Nonsustained ventricular tachycardia | 3 years
  Rate >150 bpm lasting <30 seconds
Ventricular fibrillation | 3 years
  Any duration
AF burden | 3 years
  Percentage of monitored time spent in AF rhythm, categorized as: 1) <0.05%, 2) 0.05% to 0.5%, 3) 0.5% to 5%, and 4) >5%
AF progression | 3 years
  Increase in burden in the second half of follow-up compared to the first half
Increase in NT-proBNP | 3 years
  Percentage increase in NT-proBNP between the first and last recorded value
Increase in left ventricular end-systolic diameter (LVESD) | 3 years
  Percentage increase in LVESD between the first and last echocardiography
Increase in pulmonary artery systolic pressure (PASP) | 3 years
  Percentage increase in PASP between the first and last echocardiography
Left atrial (LA) enlargement | 3 years
  LA size of >60 mL
Development of clinically diagnosed AF | 3 years
  Symptomatic AF diagnosed at an in- or out-patient contact with a 12-lead electrocardiogram with AF in its entire length or long-term heart rhythm monitoring with ≥30 sec of AF
Diagnosis of HF | 3 years
  HF diagnosed in an out-patient clinic or hospitalization for HF (criteria: HF as a primary diagnosis, admission ≥24 hours, presenting with symptoms and objectives signs and laboratory findings of HF and receiving HF treatment)
Change in symptoms and quality of life | 3 years
  Measured by changes in participant-reported HeartQol questionnaire. Minimum score 0 and maximum score 42 where a higher score indicates a better health status
Initiation, discontinuation, or adjustment of antiarrhythmic medications | 3 years
  Recorded from electronic medical records
Initiation of anticoagulation therapy | 3 years
  Recorded from electronic medical records
Referral to or performance of cardiac surgery | 3 years
  Recorded from electronic medical records
Hospitalization ≥24 hours (all-cause and cardiovascular-specific) | 3 years
  Recorded via electronic medical records Cardiovascular hospitalization: Hospitalization due to structural heart disease, worsening or de novo heart failure, arrhythmia, ischemic heart disease, venous thromboembolism, stroke.
Stroke or systemic embolism | 3 years
  Recorded via electronic medical records Criteria stroke: diagnosed in an in- or outpatient setting with new-onset focal or global neurological dysfunction lasting ≥24 hours, preferably confirmed by imaging or combined with initiation of anticoagulation therapy Criteria systemic embolism: clinical history consistent with an acute loss of blood flow in a peripheral artery with evidence of embolism (identified surgically, by autopsy or imaging)
Cardiovascular and all-cause mortality | 3 years
  Recorded via electronic medical records Cardiovascular (CV) death includes any death resulting from an acute myocardial infarction, sudden cardiac death, sudden death, death due to HF, death due to stroke, death due to CV procedures, death due to CV hemorrhage, and death due to other CV causes

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No